CLINICAL TRIAL: NCT05170360
Title: Evaluation of Some Risk Factors Associated With Colorectal Cancer and Their Correlation With KRAS and BRAF Genes Mutations
Brief Title: Evaluation of Some Risk Factors Associated With Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sarah Abdelsamee Mohammed Ali, Assistant lecturer in Forensic Medicine and Clinical Toxicology Department, Assiut University
Other Study IDs: colorectal cancer risk factors
Record Dates: First submitted 2021-12-05; First posted 2021-12-28 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The DNA will be extracted from the primary tumor tissue and adjacent noncancerous tissues using the DNA extraction kit (proteinase K and phenol extraction) and then will be stored at 4 °C, for examining the mutations in the K-ras gene and BRAF
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patient group: Patients who are recently diagnosed with CRC based on clinical and pathological examinations
  Interventions: Diagnostic Test: Assessment of smoking ,heavy metal, organophosphorus exposure and d) Mutational analysis of the KRAS and BRAF genes:
- control group: Control subjects will be CRC-free, based on the clinical history and physical examination.
  Interventions: Diagnostic Test: Assessment of smoking ,heavy metal, organophosphorus exposure and d) Mutational analysis of the KRAS and BRAF genes:

INTERVENTIONS:
Diagnostic Test: Assessment of smoking ,heavy metal, organophosphorus exposure and d) Mutational analysis of the KRAS and BRAF genes: — 1. Assessment of smoking exposure:
     Serum cotinine will be measured by using serum cotinine ELISA kits
  2. Assessment of heavy metal exposure:
     Lead and cadmium will be measured using Graphite Tube Atomizer.
  3. Assessment of organophosphorus exposure:
     By measuring pseudocholinesterase level by spectrophotometer
  4. Mutational analysis of the KRAS and BRAF genes:
  the tissue samples will be used to determine the mutation in k-ras and BRAF genes by RCR

SUMMARY:
1. Evaluation of some risk factors (e.g. smoking, heavy metal exposure, and organophosphorus exposure) on CRC.
2. Estimation of KRAS and BRAF genes mutations associated with CRC.
3. Association between different risk factors and gene mutations on different types of CRC.

DETAILED DESCRIPTION:
* Colorectal cancer (CRC) ranks as the third most common cancer globally and second in terms of mortality (Bray et al., 2018). CRC is the 7th commonest cancer in Egypt, representing 3.47% of male cancers and 3% of female cancers (Metwally et al.,2018).
* Studies have provided that rising CRC rates are associated with increased alcohol use, physical inactivity, high intake of fat, red and processed meat, and processed foods; and low intake of fiber (Zhou and Rifkin, 2021).
* Smoking is an established risk factor for colorectal adenomas as well as CRC incidence and mortality, which suggests that it may affect the prognosis of CRC patients as well (Walter et al., 2014).
* Heavy metals are natural components of the earth's crust, which, if released into the environment, can persist for many years (Wu et al., 2016). The most toxic elements are arsenic, cadmium, chromium, copper, mercury, and lead with the majority of them being classified as certainly or probably carcinogenic (Forte et al., 2020).
* Pesticides that are applied to farms can remain in the environment for longer than intended (Sjerps et al., 2019). Pesticides increase the risk of cancer through a variety of mechanisms including genotoxicity, epigenetic effects, hormonal action, and immunotoxicity (Lyons and Watterson, 2010).
* Of the key genes of CRC, KRAS mutations are the most widely known, as they are mainly localized in codons 12 and 13, which were among the first linked to the pathogenesis of colon cancer (Kudryavtseva et al., 2016). BRAF is an oncogene located on chromosome 7 for which gain of function mutations in multiple solid tumors, such as colon cancer (Frisone et al., 2020).

ELIGIBILITY:
Inclusion Criteria:

- 1. Patients who are recently diagnosed with CRC based on clinical and pathological examinations.

2. Control subjects will be CRC-free, based on the clinical history and physical examination.

Exclusion Criteria:

1 - Patient refuses to be enrolled in the study. 2. Subjects with cancer metastasized from other tissues to the colon. (colon is the site of metastasis)

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: the patient group is 50 patients who are recently diagnosed with CRC based on clinical and pathological examinations.
  THE control group is 50 subjects who will be CRC-free, based on the clinical history and physical examination.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
1. association between some risk factors and colorectal cancer | baseline
  association between smoking( by measuring serum cotinine ng/ml) , heavy metal (by measuring lead and cadmium in the blood μg/dLwill be measured using Graphite Tube Atomizer) , organophosphorus exposure (By measuring serum pseudocholinesterase level U/ml by spectrophotometer) and colorectal cancer incidience

SECONDARY OUTCOMES:
1. Estimation of KRAS and BRAF genes mutations associated with CRC. 3. Association between these risk factors and gene mutations on different types of CRC. | baseline
  Surgically resected specimens will be collected; the samples will be used to determine the mutation in k-ras and BRAF genes by PCR
  Risk factor smoking, heavy metal (lead and cadmium), organophosphorus exposure association between smoking( by measuring serum cotinine ng/ml), heavy metal (by measuring lead and cadmium in the blood μg/dLwill be measured using Graphite Tube Atomizer), organophosphorus exposure (By measuring serum pseudocholinesterase level U/ml by spectrophotometer), and colorectal cancer incidence

CONTACTS AND LOCATIONS:
Overall Officials: Hayam Z Thabet, prof.DR, Study Director — Assiut University; Heba A. Yassa, prof.DR, Study Director — Assiut University

REFERENCES:
- [Background] Erratum: Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2020 Jul;70(4):313. doi: 10.3322/caac.21609. Epub 2020 Apr 6. No abstract available. PMID 32767693
- [Background] Forte IM, Indovina P, Costa A, Iannuzzi CA, Costanzo L, Marfella A, Montagnaro S, Botti G, Bucci E, Giordano A. Blood screening for heavy metals and organic pollutants in cancer patients exposed to toxic waste in southern Italy: A pilot study. J Cell Physiol. 2020 Jun;235(6):5213-5222. doi: 10.1002/jcp.29399. Epub 2019 Dec 15. PMID 31838757
- [Background] Kudryavtseva AV, Lipatova AV, Zaretsky AR, Moskalev AA, Fedorova MS, Rasskazova AS, Shibukhova GA, Snezhkina AV, Kaprin AD, Alekseev BY, Dmitriev AA, Krasnov GS. Important molecular genetic markers of colorectal cancer. Oncotarget. 2016 Aug 16;7(33):53959-53983. doi: 10.18632/oncotarget.9796. PMID 27276710
- [Background] Nanda MS, Sameer AS, Syeed N, Shah ZA, Murtaza I, Siddiqi MA, Ali A. Genetic aberrations of the K-ras proto-oncogene in bladder cancer in Kashmiri population. Urol J. 2010 Summer;7(3):168-73. PMID 20845292
- [Background] Przybojewska B, Jagiello A, Jalmuzna P. H-RAS, K-RAS, and N-RAS gene activation in human bladder cancers. Cancer Genet Cytogenet. 2000 Aug;121(1):73-7. doi: 10.1016/s0165-4608(00)00223-5. PMID 10958945
- [Background] Frisone D, Friedlaender A, Malapelle U, Banna G, Addeo A. A BRAF new world. Crit Rev Oncol Hematol. 2020 Aug;152:103008. doi: 10.1016/j.critrevonc.2020.103008. Epub 2020 May 26. PMID 32485528
- [Background] Sjerps RMA, Kooij PJF, van Loon A, Van Wezel AP. Occurrence of pesticides in Dutch drinking water sources. Chemosphere. 2019 Nov;235:510-518. doi: 10.1016/j.chemosphere.2019.06.207. Epub 2019 Jun 27. PMID 31280041
- [Background] Walter V, Jansen L, Hoffmeister M, Brenner H. Smoking and survival of colorectal cancer patients: systematic review and meta-analysis. Ann Oncol. 2014 Aug;25(8):1517-25. doi: 10.1093/annonc/mdu040. Epub 2014 Mar 31. PMID 24692581
- [Background] Wu X, Cobbina SJ, Mao G, Xu H, Zhang Z, Yang L. A review of toxicity and mechanisms of individual and mixtures of heavy metals in the environment. Environ Sci Pollut Res Int. 2016 May;23(9):8244-59. doi: 10.1007/s11356-016-6333-x. Epub 2016 Mar 11. PMID 26965280
- [Background] Zhou E, Rifkin S. Colorectal Cancer and Diet: Risk Versus Prevention, Is Diet an Intervention? Gastroenterol Clin North Am. 2021 Mar;50(1):101-111. doi: 10.1016/j.gtc.2020.10.012. PMID 33518157